CLINICAL TRIAL: NCT02905773
Title: Postoperative Pain After the Removal of Root Canal Filling Material Using Different Techniques in Teeth With Failed Root Canal Therapy: A Randomized Clinical Trial
Brief Title: Postoperative Pain After the Removal of Root Canal Filling Material
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Hüseyin Sinan TOPÇUOĞLU, Associate Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 232/2015
Record Dates: First submitted 2016-09-06; First posted 2016-09-19 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Postoperative Pain
Keywords: Intensity
MeSH Terms: conditions — Pain, Postoperative | interventions — Root Canal Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- postoperative pain (Other): postoperative pain
  Interventions: Other: root canal therapy
- intensity (Other): intensity
  Interventions: Other: root canal retreatment

INTERVENTIONS:
Other: root canal therapy — effect of devices ( ProTaper and Reciprocal Files)
  Arms: postoperative pain
Other: root canal retreatment — effect of devices ( ProTaper and Reciprocal Files)
  Arms: intensity

SUMMARY:
The aim of this study was to evaluate the intensity and duration of postoperative pain after the removal of root canal filling material in retreatment procedures of upper incisor teeth with chronic apical periodontitis, using different techniques.

The patients were assigned to three groups of 45 patients, according to the method used to remove old canal filling material. The presence of postoperative pain was assessed after 6, 12, 24, 48, and 72 hours, 7 days, and finally after 10 days.

The hypothesis of this study: there would be no difference in postoperative pain intensity among the groups.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic incisor teeth with chronic apical periodontitis
* patients between 18-55 years of age

Exclusion Criteria:

* patients with systemic disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
postoperative pain after non-surgical endodontic retreatment using modified visual analog scale | 10 days